CLINICAL TRIAL: NCT05925413
Title: Cadonilimab Combined With Transarterial Chemoembolization (TACE) in Patients With Intermediate-stage Unresectable Hepatocellular Carcinoma: A Single Center, Single Arm, Phase II Trial
Brief Title: Cadonilimab Plus TACE in Patients With Intermediate-stage Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Professor and Chief Surgeon, Eastern Hepatobiliary Surgery Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2023-H006-P001
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+TACE (Experimental): Cadonilimab (15mg/kg Q3W D1)+TACE
  Interventions: Drug: Cadonilimab+TACE

INTERVENTIONS:
Drug: Cadonilimab+TACE — Cadonilimab: 15mg/kg Q3W Day1 Select the best TACE treatment strategy. Traditional TACE (cTACE) or DEB-TACE can be selected. TACE treatment can be continued as needed based on disease control. The combination of cadonilimab is given 3 to 7 days after the first TACE treatment, and the subsequent administration of cardonilizumab is given once every 3 weeks, if the time overlaps with TACE treatment, it is generally administered 3 to 7 days after TACE treatment. Treatment was discontinued until intolerable toxicity, death, withdrawal of informed consent, initiation of a new antitumor therapy, or other reason specified in the protocol, whichever occurs first. Patients in this study received cadonilimab for up to 24 months.

SUMMARY:
Cadonilimab is a first-in-class bispecific, humanized IgG1 antibody targeting PD-1 and CTLA-4, which has the potential to boost immune surveillance in tumors. The goal of this clinical trial is to evaluated the efficacy and safety of cadonilimab combined with TACE in patients with intermediate-stage unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent signed prior to enrolment.
2. age > 18 years, both sexes
3. patients with histologically or pathologically confirmed intermediate hepatocellular carcinoma; BCLC stage B or CNLC stage II
4. no previous antitumor therapy
5. Child-Pugh A or B7.
6. with measurable lesions (≥10 mm long diameter on CT scan for non-lymph node lesions and ≥15 mm short diameter on CT scan for lymph node lesions according to RECIST 1.1 criteria).
7. ECOG PS score: 0 to 1.
8. expected survival of >12 weeks.
9. Adequate organ function

Exclusion Criteria:

1. BCLC C stage HCC
2. In combined with severe heart, lung, kidney or other important organ dysfunction, or combined with serious infection or other serious associated diseases, that cannot tolerate treatment (> CTCAE Version 5.0 adverse events of grade 2).
3. With uncontrolled hepatitis B (HBV-DNA>2000 IU/ml and elevated ALT).
4. Multi-nodules hepatocellular carcinoma beyond hemi-hepatic range.
5. Patients with tumor thrombus reaches or exceeds the portal vein.
6. History of other malignancies.
7. History of allergic reactions to related drugs.
8. History of organ transplantation.
9. Pregnant women, nursing mothers.
10. Patients have other factors that may interfere with patient enrollment and assessment results.
11. Refuse follow-up as required by this study protocol and refuse to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year
  ORR is defined as the percentage of participants who have a confirmed complete response or partial response according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to two years
  PFS is defined as the time from enrollment of the trial to the first documented disease progression or death due to any cause.
Overall survival (OS) | Up to two years
  The duration from the date of recruitment to the date of death from any cause.
Adverse events (safety) | Up to two years
  Adverse events (safety ) will be evaluated according to the NCI CTCAE Version 5.0.The number and severity of treatment-related side effects, including AE and SAE, will be recorded during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No